CLINICAL TRIAL: NCT04862442
Title: Comparison of Qigong Exercises on Two Different Digital Platforms: an Evaluation Project of Technologically Supported Activity
Brief Title: Comparison of Qigong Exercises on Two Different Digital Platforms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Associated Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2015-KAEK-47-21-02
Record Dates: First submitted 2021-04-20; First posted 2021-04-28 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Health Behavior; Sedentary Behavior
Keywords: Qigong; telerehabilitation; physical activity
MeSH Terms: conditions — Health Behavior; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: A total of 30 volunteer research subjects will be selected in an age range of 18 to 65, who categorized as "inactive (<600 metabolic equivalent-min/hf)" with respect to International Activity Readiness Survey. Groups will be randomized as Group A (n=15) and Group B (n=15).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessors will be blind to the group allocation. The investigators will be blind to the outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1=Video-conference based Qigong exercises (Experimental): After initial result evaluation, participants of Group A will perform Qigong exercises for 40 to 45 minutes per session for 3 days a week for 6 weeks via the online video conference method.
  Interventions: Other: Qigong exercises
- Group 2=A-synchronized video Qigong exercises (Experimental): Group B will perform the same routine via a-synchronized video sections for 6 weeks.
  Basic Qigong exercises will be performed by volunteers for 6 weeks and progression will be logged.
  Interventions: Other: Qigong exercises

INTERVENTIONS:
Other: Qigong exercises — Specific Qigong exercises 1- Painting the rainbow 2-Raising the arms 3-Looking at the moon 4- Pushing the waves

SUMMARY:
Mild effort requiring, body-mind oriented, effective on multiple physical fitness parameters, ancient exercise method Qigong would be beneficial for a great number of people by using popular technological mediums in order to increase overall physical activity and wellbeing. Our aim is to evaluate the effects of Qigong exercises on endurance, muscle strength, sleep quality, level of anxiety and stress by using two different tele-rehabilitation methods.

DETAILED DESCRIPTION:
Physical inactivity and sedentary behavior is a serious public health problem which categorized as a pandemic. One of the common risk factors for cardiovascular diseases, cancers, chronic respiratory diseases and diabetes, known as chronic non-communicable diseases, is physical inactivity. Mild effort requiring, body-mind oriented, effective on multiple physical fitness parameters, ancient exercise method Qigong would be beneficial for a great number of people by using popular technological mediums in order to increase overall physical activity and wellbeing. Based on reasons as previously described, our aim is to evaluate the effects of Qigong exercises on endurance, muscle strength, sleep quality, level of anxiety and stress by using two different tele-rehabilitation methods.

ELIGIBILITY:
Inclusion Criteria:

* • Categorized as "inactive (<600 metabolic equivalent-min/hf)" with respect to International Physical Activity Questionnaire

  * Ability to read and talk in Turkish
  * In order to join online sessions, participants should have internet access
  * All answers of the Physical Activity Preparation Survey should be selected as "No"

Exclusion Criteria:

* • Lack of cooperation

  * Uncontrolled hypertension and uncontrolled arrhythmia patience
  * People with serious neurological and respiratory conditions
  * Having a pacemaker and/or percutaneous transluminal coronary angioplasty
  * Stroke, myocardial infarction history
  * Amputee
  * People with serious major musculoskeletal problems
  * Chronic kidney failure
  * Chronic Liver failure
  * Hip or knee prosthesis in last five years
  * Lower extremity injuries in last 6 months
  * Diabetic ulcer or neuropathy
  * Pregnant or planning to get pregnant in 1 year
  * Breastfeeding
  * Taking sleep pills or taking medicines as part of psychological treatment and/or working on shifts

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire-Short form | 8 weeks
  Determines the physical activity level of the participants

SECONDARY OUTCOMES:
1 Minute Sit-Stand Test | 8 weeks
  Determines the functional mobility and lower extremity levels
Pittsburgh Sleep Quality Index | 8 weeks
  Determines the sleep quality of participants
Coronavirus Anxiety Index | 8 weeks
  Determines the coronavirus anxiety
Perceived Stress Index | 8 weeks
  Determines the perceived stress

CONTACTS AND LOCATIONS:
Overall Officials: Buket Akinci, Assoc.Prof., Study Chair — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared